CLINICAL TRIAL: NCT04631614
Title: Addition Effect of the Calf Stretching and Ankle Mobilization to Quadriceps and Gluteus Strengthening on Knee Pain and Function in Women With Patellofemoral Pain: a Randomized Controlled Trial
Brief Title: Addition Effect of the Ankle Manual Therapy to Muscle Strengthening Exercise in Women With Patellofemoral Pain
Acronym: PhD_Bruno
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Gabriel Peixoto Leão Almeida, Professor, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PhD_Bruno
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: knee; pain; ankle; manual therapy; exercise
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain; Motor Activity | interventions — Warm-Up Exercise; Movement; Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy plus muscle strengthening exercises (Experimental): The procedures to be performed with participants in the experimental group are as follows: (1) warm up with a walk or exercise bike for 5 minutes; (2) two ankle manual therapy techniques - [a] passive calf muscle stretching and [b] ankle joint mobilization; (3) five muscle strengthening exercises focusing on quadriceps and posterolateral hip complex - [a] clam exercise, [b] hip abduction exercise in side lying, [c] knee extension exercise in a sitting position, [d] squat exercise and [e] forward lunge exercise.
  Interventions: Other: Warm up; Other: Passive calf muscle stretching; Other: Ankle joint mobilization - weight-bearing mobilization with movement (WB-MWM) technique; Other: Clam exercise; Other: Hip abduction exercise in side lying; Other: Knee extension exercise in a sitting position; Other: Squat exercise; Other: Forward lunge exercise
- Muscle strengthening exercises (Active Comparator): The procedures to be performed with participants in the control group are as follows: (1) warm up with a walk or exercise bike for 5 minutes; (2) five muscle strengthening exercises focusing on quadriceps and posterolateral hip complex - [a] clam exercise, [b] hip abduction exercise in side lying, [c] knee extension exercise in a sitting position, [d] squat exercise and [e] forward lunge exercise.
  Interventions: Other: Warm up; Other: Clam exercise; Other: Hip abduction exercise in side lying; Other: Knee extension exercise in a sitting position; Other: Squat exercise; Other: Forward lunge exercise

INTERVENTIONS:
Other: Warm up — Warm up through a walk or exercise bike for 5 minutes with moderate intensity according to modified Borg scale (CR-10)
Other: Passive calf muscle stretching — With the participant lying in the supine position, the physiotherapist will passively perform the ankle dorsiflexion movement to stretch the participant's calf to the limit tolerated by the participant. This procedure will be performed in two repetitions with 30 seconds of held in the stretching position and 30 seconds of rest between repetitions.
  Arms: Manual therapy plus muscle strengthening exercises
Other: Ankle joint mobilization - weight-bearing mobilization with movement (WB-MWM) technique — To perform the WB-MWM technique, the participant will be instructed to take a weight-bearing position with the tibia in a vertical position. The physiotherapist will be stay in front participant's ankle and will use the hands to stabilize the participant's foot as close as possible to the anterior region of the talus. A rigid belt will be placed on the participant's tibia and around physiotherapist´s hip. Then, the physiotherapist will project his hip backwards to produce a nonpainful anterior tibia glide. The participant will be asked to perform a forward lunge as far as possible without raising heel off the table and without reproducing knee symptoms. After achieving the maximum forward lunge, the participant will be instructed to hold this position for 5 seconds and then return to the starting position. This procedure will be performed in two sets of 10 repetitions with two minutes of rest between sets.
  Arms: Manual therapy plus muscle strengthening exercises
Other: Clam exercise — The participant will side lying with trunk straight and both hips and knees at 45º and 90º of flexion, respectively. An elastic band will be used as external resistance, that will be positioned above the participant's knee. The individual will be instructed to perform the abduction and lateral rotation of the hip (keeping the heels in contact) against the resistance of the elastic band and then return to starting position. This exercise will be performed in three sets of 12 repetitions with on minutes of rest between sets. The exercise will be carried out with a load between 60-80% of the capacity and level of effort reported by the participant, according to the specifications of the modified Borg scale (CR-10). The load will be increased by 2-10% when the patient is able to perform 12 full repetitions in the last set of the exercise with perceived effort <60%.
Other: Hip abduction exercise in side lying — The participant will side lying with trunk straight, both hips in a neutral position and both knee in extension. An elastic band will be used as external resistance, that will be positioned above the participant's knee. The individual will be instructed to perform the hip abduction against the resistance of the elastic band and then return to starting position. This exercise will be performed in three sets of 12 repetitions with with on minutes of rest between sets. The exercise will be carried out with a load between 60-80% of the capacity and level of effort reported by the participant, according to the specifications of the modified Borg scale (CR-10). The load will be increased by 2-10% when the patient is able to perform 12 full repetitions in the last set of the exercise with perceived effort <60%.
Other: Knee extension exercise in a sitting position — The participant will be seated at the treatment table with the trunk straight and both knees in 90º of flexion. The external resistance will be positioned above the participant's ankle. The individual will be instructed to perform the knee extension at a protective angle (90º-45º of flexion), progressing to full extension (90º-0º of flexion) as long as the full knee extension does not reproduce the knee pain symptoms. Then, the participant will should return to starting position. This exercise will be performed in three sets of 12 repetitions with with on minutes of rest between sets. The exercise will be carried out with a load between 60-80% of the capacity and level of effort reported by the participant, according to the specifications of the modified Borg scale (CR-10). The load will be increased by 2-10% when the patient is able to perform 12 full repetitions in the last set of the exercise with perceived effort <60%.
Other: Squat exercise — The participant will be stand with the trunk straight, knees in extension and feet hip-width apart. Dumbbells will be used as external resistance.The individual will be instructed to perform the squat movement at a protective angle (0º-45º of knee flexion), progressing to a deep squat (90º of knee flexion) as long as the movement does not reproduce the knee pain symptoms. Then, the participant will should return to starting position. This exercise will be performed in three sets of 12 repetitions with with on minutes of rest between sets. The exercise will be carried out with a load between 60-80% of the capacity and level of effort reported by the participant, according to the specifications of the modified Borg scale (CR-10). The load will be increased by 2-10% when the patient is able to perform 12 full repetitions in the last set of the exercise with perceived effort <60%.
Other: Forward lunge exercise — The participant will be stand with one lower limb in a long stride forwards of the other limb, trunk straight and both knee in extension. Dumbbells will be used as external resistance. From this position, the participant will be instructed to bend both knees to lower your body at a protective angle (0º-45º of knee flexion), progressing to a greater knee flexion (90º) as long as the movement does not reproduce the knee pain symptoms. Then, the participant will should return to starting position. This exercise will be performed in three sets of 12 repetitions with with on minutes of rest between sets. The exercise will be carried out with a load between 60-80% of the capacity and level of effort reported by the participant, according to the specifications of the modified Borg scale (CR-10). The load will be increased by 2-10% when the patient is able to perform 12 full repetitions in the last set of the exercise with perceived effort <60%.

SUMMARY:
Patellofemoral pain (PFP) is the most common overuse injury of the lower limb, its prevalence is around 20% in general population, and women are more likely to develop PFP compared to men. PFP may develop as a result of increased pressure and joint stress due to an reduction in contact area in the patellofemoral joint. The excessive dynamic knee valgus is an important contributor to patella misalignment and for the increasing of laterally directed forces on the patella, and restriction in ankle dorsiflexion range of motion (ROM) has been previously associated with excessive dynamic knee valgus. Although the evidence shows that strengthening exercises for the quadriceps and gluteus promote improvement of knee pain and function, there is a lack of studies that investigate if targeted interventions for improvement ankle dorsiflexion may promote additional benefits in knee pain and function when performed in combination with strengthening exercises. Thus, the aimed of this study is analyze the addition effect of calf stretching and ankle mobilization to quadriceps and gluteus strengthening on knee pain and function in women with PFP who display ankle dorsiflexion restriction.

DETAILED DESCRIPTION:
The study sample will be formed by 68 women with PFP who show ankle dorsiflexion restriction, divided into two groups: Experimental Group (EG, n = 34), that will receive two manual therapy techniques (calf muscle stretching and ankle mobilization) followed by five muscle strengthening exercises focusing on quadriceps and posterolateral hip complex (PHC), and; Control Group (CG, n = 34), that will receive only the five muscle strengthening exercises focusing on quadriceps and PHC. The treatment sessions will be individual and supervised by a physiotherapist, will last 40-50 minutes and will perform twice a week for six weeks. Before starting each treatment session, both groups will perform warm up with a walk or exercise bike for 5 minutes.

The calf muscle stretching will be performed passively in two repetitions with 30 seconds of held in the stretching position and 30 seconds of rest between repetitions. The ankle mobilization will be performed using the Weight-bearing Mobilization with Movement (WB-MWM) technique, being applied in two sets of 10 repetitions with two minutes of rest between sets.

The five muscle strengthening exercises will be as follows: (a) clam exercise; (b) hip abduction exercise in side lying; (c) knee extension exercise in a sitting position; (d) squat exercise, and; (e) forward lunge exercise. All exercises will be performed in three sets of 12 repetitions with on minutes of rest between sets and two minutes of rest between exercises.

Regarding the intensity of the exercises, this will be monitored by the physiotherapist according to the perception of the level of effort and difficulty reported by the participant when completing the series of each exercise, according to the specifications of the modified Borg scale (CR-10). The exercises will be carried out with a load between 60-80% of the capacity and level of effort reported by the participant. The load will be increased by 2-10% when the patient is able to perform 12 full repetitions in the last series of the exercise with perceived effort <60%.

ELIGIBILITY:
Inclusion Criteria:

* Presence of anterior knee pain for at least 3 months, unrelated to any traumatic knee event and reproducible by performing at least two of the following activities: sitting for a long time, squatting, kneeling, ascending or descending stairs, walking or running long distances, and performing jump-landing tasks;
* Anterior knee pain in the previous week with an intensity of at least 3 points on numeric pain rating scale (NPRS);
* Score in the Anterior Knee Pain Scale less than or equal to 86 points, and;
* Limited ankle dorsiflexion range of motion in closed kinetic chain, identified by a weight-bearing lunge test in which the distance between foot and wall being less than or equal to 10 cm.

Exclusion Criteria:

* History of surgery or fracture in the lumbar spine, hip, knee, ankle, or foot;
* Referred pain from the lumbar spine, hip, ankle, or foot;
* History of patellar subluxation;
* Presence of knee swelling;
* Presence of meniscal, ligament or tendon injury, and;
* Osgood-Schlatter or Siding-Larsen-Johansson syndrome.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | At the end of the six weeks of treatment
  Pain will be assessed by use of an 11-point Numeric Pain Scale, where 0 correspond to no pain and 10 correspond to worst imaginable pain.
Anterior Knee Pain Scale | At the end of the six weeks of treatment
  The subjective functional capacity of the participant will be recorded with the translated and validated Portuguese-language version of the Anterior Knee Pain Scale (AKPS). The scores for this scale, 0 to 100, represent the lowest to the highest levels of functional capacity, respectively.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | At 3 and 6 months follow-up
  Pain will be assessed by use of an 11-point Numeric Pain Scale, where 0 correspond to no pain and 10 correspond to worst imaginable pain.
Anterior Knee Pain Scale | At 3 and 6 months follow-up
  The subjective functional capacity of the participant will be recorded with the translated and validated Portuguese-language version of the Anterior Knee Pain Scale (AKPS). The scores for this scale, 0 to 100, represent the lowest to the highest levels of functional capacity, respectively.
Weight-Bearing Lunge Test | At the end of the six weeks of treatment
  The ankle dorsiflexion range of motion in closed kinetic chain will be measured by the distance between foot and wall in the weight-bearing lunge test.
Dynamic knee valgus | At the end of the six weeks of treatment
  The dynamic knee valgus will be assessed by 2D kinematic through measurement of frontal plane projection angle of the knee during the forward step-down test.
Isometric strength of the quadriceps | At the end of the six weeks of treatment.
  The quadriceps isometric strength will be assessed using a handheld dynamometer (Nicholas Manual Muscle Test, Lafayette Instrument Company, Lafayette, Indiana, USA). The evaluation will be performed with the participant in a sitting position, straight trunk and knee at 90º of flexion.
Isometric strength of the hip posterolateral complex | At the end of the six weeks of treatment.
  The hip posterolateral complex isometric strength will be assessed using a handheld dynamometer (Nicholas Manual Muscle Test, Lafayette Instrument Company, Lafayette, Indiana, USA) during the Hip Stability Isometric Test (HipSIT).
Global Effect Perception Scale for Treatment | At the end of the six weeks of treatment.
  The participant's perception of treatment will be assessed by use of an 11-point Global Effect Perception Scale , where +5 correspond to perception of great improvement and -5 correspond to perception of great worsening.

CONTACTS AND LOCATIONS:
Locations (1):
- Bruno Augusto Lima Coelho, Fortaleza, Ceará, Brazil